CLINICAL TRIAL: NCT05228145
Title: A Phase 1/2 Intracerebroventricular and Intravitreal Administration of NGN-101 for Treatment of Neuronal Ceroid Lipofuscinosis (NCL) Subtype 5 (CLN5) Disease
Brief Title: Gene Therapy Study for Children With CLN5 Batten Disease
Acronym: CLN5-200
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neurogene Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN5-200
Record Dates: First submitted 2021-12-17; First posted 2022-02-08 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Neuronal Ceroid Lipofuscinosis CLN5
Keywords: Batten Disease; Neuronal Ceroid Lipofuscinosis Disease; Neuronal Ceroid Lipofuscinosis Subtype 5 Disease; NCL; Gene Therapy; Gene Transfer; CLN5; CLN
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Intervention Model Description: Dose escalation cohort study of NGN-101 administered by intracerebroventricular (ICV) infusion and intravitreal (IVT) injection; cohorts will be assigned sequentially.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): The study treatment is a recombinant serotype 9 adeno-associated virus encoding a codon-optimized human CLN5 transgene (hCLN5opt).
  Interventions: Genetic: NGN-101
- Cohort 2 (Experimental): The study treatment is a higher dose of recombinant serotype 9 adeno-associated virus encoding a codon-optimized human CLN5 transgene (hCLN5opt).
  Interventions: Genetic: NGN-101
- Cohort 3 (Experimental): The study treatment is a higher dose of recombinant serotype 9 adeno-associated virus encoding a codon- optimized human CLN5 transgene (hCLN5opt).
  Interventions: Genetic: NGN-101

INTERVENTIONS:
Genetic: NGN-101 — Participants with confirmed mutations in the CLN5 gene who meet all the inclusion and none of the exclusion criteria will be treated with a single intracerebroventricular (ICV) dose and a single intravitreal (IVT) dose of the study treatment.

SUMMARY:
This is a prospective, non-randomized, open-label, dose escalation study of a single administration of gene therapy in children who are 3 to 9 years old with Neuronal Ceroid Lipofuscinosis (Batten) Subtype 5 (CLN5) disease.

DETAILED DESCRIPTION:
The study is a first in human (FIH) open-label, dose escalation study designed to assess the safety and efficacy of administration of an adeno-associated viral vector serotype 9 (AAV9) carrying the gene encoding human ceroid-lipofuscinosis neuronal protein 5 (CLN5) in subjects with CLN5 Batten disease. The study treatment will be delivered via intracerebroventricular (ICV) and intravitreal (IVT) injection on the same day. Each participant will be followed for safety and efficacy for 5 years after treatment. Efficacy assessments in this study will evaluate motor, language, visual and cognitive function.

ELIGIBILITY:
Inclusion Criteria

* Age from 3 to 9 years (Child)
* Molecular genetic diagnosis of the CLN5 gene
* Confirmed clinical diagnosis of CLN5 disease
* Impaired motor and/or language function and/or impaired visual acuity
* Written informed consent from parent or legal guardian and assent from study participant, if appropriate
* Able to comply with protocol required assessments (laboratory sample collection, lumbar puncture (LP), nerve conduction studies (NCS), magnetic resonance imaging (MRI), etc.), which may require sedation or general anesthesia
* Able to walk with or without assistance (assistance may include a walker, braces, or with one hand held)
* Agree to reside within a 1-hour drive of the study site for at least 6 months following treatment (or a safely drivable distance for the study participant and caregivers according to investigator's discretion)

Exclusion Criteria

* Has another neurologic disease or illness that may have caused cognitive decline before study entry
* Known pathogenic or clinically suspected variant in a seizure associated genetic mutation besides CLN5
* Any active infections or severe infections within the 30 days prior to study treatment administration
* Presence of a concomitant medical condition that precludes intracerebroventricular (ICV) injection, lumbar puncture (LP), or use of anesthetics needed for study-related procedures
* Presence of any concomitant medical conditions that preclude intravitreal (IVT) administration
* Has status epilepticus that lasts longer than 5 minutes or having more than 1 seizure within a 5-minute period, without returning to a normal level of consciousness between episodes within 12 weeks before study treatment
* Total anti-AAV9 antibody titer greater than 1:400
* Any anticipated need for major surgery in the next 24 months
* Participation in an Investigational New Drug, Investigational Device Exemption, or equivalent clinical study in the past 6 months
* Any prior participation in a study in which a gene therapy vector or stem cell transplantation was administered
* Participation in other investigational studies and non-interventional studies that have similar study assessments as this protocol while the study participant is enrolled in this study with the exception of sister studies sponsored by Neurogene
* History of or current chemotherapy, radiotherapy, or other immunosuppressive therapy within the past 3 months
* Use of prohibited medications
* Immunizations of any kind in the 45 days prior to study treatment
* Requiring daytime or nighttime ventilatory support at the time of Screening
* Any item which would exclude the study participant from being able to undergo brain magnetic resonance imaging (MRI) according to local institutional policy
* Known allergies or hypersensitivities to the required immunosuppression regime

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | 5 years (multiple visits)
  Incidence, type, severity, and frequency of TEAEs
Incidence of Serious Adverse Events (SAEs) | 5 years (multiple visits)
  Incidence, type, severity, and frequency of SAEs
Incidence of clinical laboratory abnormalities | 5 years (multiple visits)
  Incidence, type, severity, and frequency of clinical laboratory abnormalities
Incidence of new nerve conduction study (NCS) abnormalities | 5 years (multiple visits)
  Incidence, type, severity, and frequency of new nerve conduction study (NCS) abnormalities
Incidence of new physical and neurologic exam abnormalities | 5 years (multiple visits)
  Incidence, type, severity, and frequency of new physical and neurologic exam abnormalities

SECONDARY OUTCOMES:
Change in Hamburg Scale, Motor and Language domain scores | 5 years (multiple visits)
  Change from baseline in Hamburg Scale, Motor and Language domain scores (each domain is rated from 0 to 3, with 3 reflecting normal function for age and 0 reflecting complete loss of function)
Change in Spectral Domain-Optical Coherence Tomography (SD-OCT) | 5 years (multiple visits)
  Change from baseline in SD-OCT parameters including Ellipsoid Zone (EZ) defect area measurements, macular volume and thickness, retinal nerve fiber layer thickness, and ganglion cell layer thickness
Change in Unified Batten Diseases Rating Scale (UBDRS) | 5 years (multiple visits)
  Change from baseline in total score and individual domains of the Unified Batten Diseases Rating Scale (UBDRS; total score 0 to 277, with higher scores indicating worse function)
Change in Caregiver global impression of change | 5 years (multiple visits)
  Caregiver global impression of change throughout the study
Change in visual acuity measurements | 5 years (multiple visits)
  Change from baseline in visual acuity measured using Teller acuity cards, Lea symbol chart, Landolt C chart, or low contrast visual acuity (measure to be used will depend on subject's level of cognitive and visual function)
Change in color vision | 5 years (multiple visits)
  Change from baseline in color vision measured using Ishihara color blindness testing

CONTACTS AND LOCATIONS:
Overall Officials: Effie Albanis, MD, Study Director — Neurogene Inc.
Locations (2):
- University of Rochester, Rochester, New York, United States
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murray SJ, Wellby MP, Barrell GK, Russell KN, Deane AR, Wynyard JR, Gray SJ, Palmer DN, Mitchell NL. Efficacy of dual intracerebroventricular and intravitreal CLN5 gene therapy in sheep prompts the first clinical trial to treat CLN5 Batten disease. Front Pharmacol. 2023 Oct 24;14:1212235. doi: 10.3389/fphar.2023.1212235. eCollection 2023. PMID 37942487
- [Derived] Mitchell NL, Murray SJ, Wellby MP, Barrell GK, Russell KN, Deane AR, Wynyard JR, Palmer MJ, Pulickan A, Prendergast PM, Casy W, Gray SJ, Palmer DN. Long-term safety and dose escalation of intracerebroventricular CLN5 gene therapy in sheep supports clinical translation for CLN5 Batten disease. Front Genet. 2023 Aug 8;14:1212228. doi: 10.3389/fgene.2023.1212228. eCollection 2023. PMID 37614821